CLINICAL TRIAL: NCT03868774
Title: The Antidepressant Effect of Right Prefrontal Low Frequency rTMS in an Accelerated Treatment Model ( rTMS). An Open Controlled, Randomized Study
Brief Title: The Antidepressant Effect of Right Prefrontal Low Frequency rTMS in an Accelerated Treatment Model
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of ressources
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Poul Erik Buchholtz, senior researcher, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADA
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: treatment
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: comparing the antidepressant effect of a standard rTMS model with an accelerated treatment model
Who Masked: Investigator, Outcomes Assessor
Masking Description: Project collaborators examining the degree of depression during intervention are blinded to the type of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS standard (Active Comparator): Low frequency (1 Hz), rTMS 20 sessions given on 20 consecutive days ( except weekends)
  Interventions: Procedure: repetitive transcranial magnetic stimulation
- rTMS accelerated model (Active Comparator): Low frequency ( 1 Hz), right prefrontal transcranial magnetic stimulation. 20 sessions given on 5 consecutive days ( 4 sessions each day)
  Interventions: Procedure: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Procedure: repetitive transcranial magnetic stimulation — rTMS is a new non-invasive antidepressant method, which implies non-convulsive focal stimulation of the prefrontal cortex of the brain through a time varying magnetic field.

SUMMARY:
Repetitive transcranial magnetic stimulation has appeared a new non-invasive antidepressant method, which implies non-convulsive focal stimulation of the prefrontal cortex of the brain through a time varying magnetic field. The method is associated with minimal side effects limited to local discomfort and especially no impact on cognitive function. The method has been approved for the treatment of depression in Canada, USA and a couple of European countries. The department for Affective Disorders, Aarhus University Hospital has used rTMS as add-on to conventional antidepressant treatment in the outpatient clinic since 2015. A single treatment course covers 20 sessions given on 20 consecutive days. The demand for daily treatment and attendance for 20 days is resource demanding for both the patient and the clinic. In consequence the investigators want to examine the antidepressant effect of an accelerated stimulus model comparing the outcome of the standard model ( 20 days) with a treatment model covering the same number of stimuli given within one week.

DETAILED DESCRIPTION:
rTMS has appeared a potential new non-invasive antidepressant method, which implies nonconvulsive focal stimulation of the brain through a time varying magnetic field. RTMS is based on the principle of electromagnetism. An electromagnetic coil placed on the scalp produces a time-varying magnetic field that penetrates the scalp and skull unattenuated and gives rise to a current in the proximity of the cerebral cortex as well as functionally connected parts of the brain. Research on rTMS reports of minimal side effects of the method.

Previous research indicates that the antidepressant effect of rTMS is associated with specific stimulation of the dorsolateral prefrontal cortex. The stimulus frequency has shown to play a key role in the mechanisms of action of rTMS. Previous animal studies have shown that low frequency rTMS is associated with long term inhibition of neuronal activity (long term depression), while high frequency stimulation is followed by prolonged activation (long term potentiation). The majority of clinically controlled studies have used high frequency stimulation of the left frontal cortex, which has been approved by the USA and later in the European Union for the treatment of depression. Fewer studies have used right prefrontal low frequency rTMS, which has less side effects, such as local discomfort and a lower risk of releasing epileptic seizures, than high frequency stimulation. Randomized controlled trials and meta-analysis have shown that both stimulus models have a clinically, significant antidepressant effect at the same level as antidepressant drugs, and recent research clearly indicates that low frequency rTMS of the right prefrontal cortex is associated with an antidepressant effect at the same level as the high frequency model. The issue indicates that low frequency due to the more advantageous side effect profile should be the stimulus model of choice in a clinical setting.

The Department for Affective Disorders, Aarhus University Hospital has taken part in rTMS research since 1999, and the outpatient clinic has used low frequency rTMS as add-on to conventional antidepressant treatment since 2015. A single treatment course covers 20 treatment sessions given on 20 consecutive days. The demand for daily treatment and attendance in the outpatient clinic for 20 days is resource demanding both for the patient and the clinic. In consequence the investigators want to examine the antidepressant effect of an accelerated stimulus model comparing the antidepressant efficacy of conventional treatment (20 days) with a treatment model covering the same number of stimuli given within one week.The study is lightening the significance of the association between the number of stimulus pulses, the length of the total treatment period and the antidepressant effect. Patients suffering for depression may benefit from the outcome of the study by obtaining an accelerated antidepressant effect from a less time consuming stimulus model. The outcome of the study may be implemented in clinical practice from day one.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate-severe uni- and bipolar depression according to the International Classification of Diseases (ICD-10)
2. A Hamilton scale score (HDS-17) of ≥ 18 and/or a sub-scale (HDSS) score of ≥ 9 within 24-48 hours before the first treatment

Exclusion Criteria:

1. Organic brain disease.
2. Epileptic seizure < 2 years
3. Patients with implanted metal parts in the brain or chest
4. Patients with pacemaker
5. Medical diseases with cerebral impact
6. Serious suicidal danger

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The Hamilton 17 item scale score for depression | up to 4 weeks
  A semistructured interview. On the basis of a systematic registration of well defined depressive symptoms through the preceding 3 days a total 17 item score and af 6-item subscale score expressing the degree of depression is calculated. The score is positively correlated to the degree af depression, Remission is defined as a total score after termination of treatment of >= 8, response is defined by >= 50% decrease in the total 17 item score during the treatment period

SECONDARY OUTCOMES:
cognitive function | 1 and 4 weeks
  Neuropsychological test of cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: Poul Erik Buchholtz, MD, Principal Investigator — Department of Depression and Anxiety

IPD SHARING:
Plan to Share IPD: No